CLINICAL TRIAL: NCT05280626
Title: First-line Treatment of P53 Mutation With PD-L1 Expression in DLBCL With Anti-PD-1 Mab and R-CHOP: a Randomized, Open, Multicenter Clinical Study
Brief Title: First-line Treatment of P53 Mutation With PD-L1 Expression in DLBCL With Anti-PD-1 Mab and R-CHOP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, sunxiuhua, Chief physician, Innovent Biologics (Suzhou) Co. Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308Y047
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — sintilimab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; Rituximab

STUDY DESIGN:
Intervention Model Description: Patients with P53 mutation with PD-L1 expressing DLBCL were randomized 1:1 into 2 groups: Group A Sindilizumab + R-CHOP and Group B R-CHOP, Sindilizumab was administered on day 10 after chemotherapy to avoid interference from prednisone. after 6 cycles, the treatment effective in Group A was maintained with Sindilizumab for 6 months as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: PD-1+R-CHOP (Experimental): After one cycle of standard R-CHOP chemotherapy, Group A uses Sindilizumab + R-CHOP, with Sindilizumab administered on day 10 post-chemotherapy, scheduled for 5 cycles. After 5 cycles, CR patients in group A continue Sindilizumab treatment for 8 times, once every 21 days.
  Interventions: Drug: Sintilimab; Drug: Rituximab
- B: R-CHOP (Active Comparator): After one cycle of standard R-CHOP chemotherapy, Group B uses R-CHOP and plans for 5 cycles. CR patients in group B are followed up for observation.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Sintilimab — After one cycle of standard R-CHOP chemotherapy, Group A uses Sintilimab with R-CHOP, with Sintilimab administered on day 10 post-chemotherapy, scheduled for 5 cycles. After 5 cycles CR patients in group A continue Sindilizumab treatment for 8 times, once every 21 days.
  Other Names: Cyclophosphamide; Doxorubicin; Oncovin; Prednisolone
  Arms: A: PD-1+R-CHOP
Drug: Rituximab — After one cycle of standard R-CHOP chemotherapy, Group B uses R-CHOP for 5 cycles. After 5 cycles, CR patients in group B are followed up for observation.
  Other Names: Cyclophosphamide; Doxorubicin; Oncovin; Prednisolone

SUMMARY:
Diffuse large B-cell lymphoma (DLBCL) is the most common type of lymphoma。The majority of refractory patients have PD-L1 expression due to P53 mutations, some of which account for about 10% of DLBCL.Our department has found that in refractory DLBCL with high PD-L1 expression, cedilizumab monotherapy is also more effective and has reversed chemotherapy resistance.The aim of this study was to determine whether the addition of sindilizumab to the R-CHOP regimen could improve the objective efficiency of DLBCL patients with P53 mutation with PD-L1 expression and to see if it could prolong patient survival.

DETAILED DESCRIPTION:
This study is a randomized, open, multicenter clinical study to determine whether the addition of sindilizumab to the R-CHOP regimen could improve the objective efficiency of DLBCL patients with P53 mutation with PD-L1 expression and to see if it could prolong patient survival.In this study, patients with P53 mutation with PD-L1 expressing DLBCL were selected to be randomised 1:1 into 2 groups: group A Sindilizumab + R-CHOP and group B R-CHOP. Sindilizumab was administered on day 10 after chemotherapy to avoid interference from prednisone.At the end of 6 cycles, Group A treatment effective maintenance treatment with Sindilizumab for 6 months as indicated.Each patient's tumour tissue was tested for mutations and ctDNA after allocation, and ctDNA and peripheral blood free PD-L1 levels were monitored dynamically during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ages≥18 years, ≤ 80 years.
2. Patients with primary treatment of DLBCL.
3. Histopathologically confirmed diagnosis of diffuse large B-cell lymphoma.
4. At least one measurable lesion according to the 2014 Lugano criteria.
5. ECOG physical status score of 0, 1 or 2.
6. Laboratory tests meet the following criteria unless judged to be due to lymphoma:

   1. Routine blood tests: (in the absence of growth factor support therapy or blood transfusion within 7 days) haemoglobin ≥ 90 g/L, absolute neutrophil value ≥ 1.5 x 109/L, platelet count ≥ 90 x 109/L.
   2. Liver biochemistry: serum creatinine ≤ 1.5 x upper limit of normal; total bilirubin ≤ 1.5 x upper limit of normal; glutamate transaminase and glutamic oxalacetic transaminase ≤ 2.5 x upper limit of normal.
   3. Coagulation: INR and APTT ≤ 2.5 times the upper limit of normal values.
7. Consent to use contraception during the trial and for 3 months after its completion.
8. Expected survival ≥ 3 months.

Exclusion Criteria:

1. Suffering from other untreated malignant tumours.
2. Cardiovascular disease that remains unstable under pharmacological control .
3. With severe interstitial lung disease.
4. With cognitive impairment.
5. Patients with uncontrolled autoimmune disease.
6. Presence of uncontrolled active infection.
7. Expected survival time < 3 months.
8. Lactating women and subjects of childbearing age who do not wish to use contraception.
9. With poor adherence or unable to follow up regularly.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CRR | 1 year
  To assess complete response rate (CRR)

SECONDARY OUTCOMES:
PFS | 1 year
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first).
ORR | 1 year
  Objective response rate (ORR)
OS | 1 year
  Defined as the time from the start of treatment to the death of the subject due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuhua Sun, Master, Principal Investigator — The Second Affiliated Hospital of Dalian Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coiffier B, Thieblemont C, Van Den Neste E, Lepeu G, Plantier I, Castaigne S, Lefort S, Marit G, Macro M, Sebban C, Belhadj K, Bordessoule D, Ferme C, Tilly H. Long-term outcome of patients in the LNH-98.5 trial, the first randomized study comparing rituximab-CHOP to standard CHOP chemotherapy in DLBCL patients: a study by the Groupe d'Etudes des Lymphomes de l'Adulte. Blood. 2010 Sep 23;116(12):2040-5. doi: 10.1182/blood-2010-03-276246. Epub 2010 Jun 14. PMID 20548096
- [Result] Young KH, Leroy K, Moller MB, Colleoni GW, Sanchez-Beato M, Kerbauy FR, Haioun C, Eickhoff JC, Young AH, Gaulard P, Piris MA, Oberley TD, Rehrauer WM, Kahl BS, Malter JS, Campo E, Delabie J, Gascoyne RD, Rosenwald A, Rimsza L, Huang J, Braziel RM, Jaffe ES, Wilson WH, Staudt LM, Vose JM, Chan WC, Weisenburger DD, Greiner TC. Structural profiles of TP53 gene mutations predict clinical outcome in diffuse large B-cell lymphoma: an international collaborative study. Blood. 2008 Oct 15;112(8):3088-98. doi: 10.1182/blood-2008-01-129783. Epub 2008 Jun 17. PMID 18559976
- [Result] McDermott DF, Atkins MB. PD-1 as a potential target in cancer therapy. Cancer Med. 2013 Oct;2(5):662-73. doi: 10.1002/cam4.106. Epub 2013 Jul 21. PMID 24403232
- [Result] Ansell SM, Minnema MC, Johnson P, Timmerman JM, Armand P, Shipp MA, Rodig SJ, Ligon AH, Roemer MGM, Reddy N, Cohen JB, Assouline S, Poon M, Sharma M, Kato K, Samakoglu S, Sumbul A, Grigg A. Nivolumab for Relapsed/Refractory Diffuse Large B-Cell Lymphoma in Patients Ineligible for or Having Failed Autologous Transplantation: A Single-Arm, Phase II Study. J Clin Oncol. 2019 Feb 20;37(6):481-489. doi: 10.1200/JCO.18.00766. Epub 2019 Jan 8. PMID 30620669
- [Result] McCord R, Bolen CR, Koeppen H, Kadel EE 3rd, Oestergaard MZ, Nielsen T, Sehn LH, Venstrom JM. PD-L1 and tumor-associated macrophages in de novo DLBCL. Blood Adv. 2019 Feb 26;3(4):531-540. doi: 10.1182/bloodadvances.2018020602. PMID 30770362
- [Result] Pascual M, Mena-Varas M, Robles EF, Garcia-Barchino MJ, Panizo C, Hervas-Stubbs S, Alignani D, Sagardoy A, Martinez-Ferrandis JI, Bunting KL, Meier S, Sagaert X, Bagnara D, Guruceaga E, Blanco O, Celay J, Martinez-Baztan A, Casares N, Lasarte JJ, MacCarthy T, Melnick A, Martinez-Climent JA, Roa S. PD-1/PD-L1 immune checkpoint and p53 loss facilitate tumor progression in activated B-cell diffuse large B-cell lymphomas. Blood. 2019 May 30;133(22):2401-2412. doi: 10.1182/blood.2018889931. Epub 2019 Apr 11. PMID 30975638